CLINICAL TRIAL: NCT04191993
Title: A Prospective Randomised Controlled Trial Comparing the Direct Superior Approach Versus the Posterior Approach for Total Hip Arthroplasty
Brief Title: Direct Superior Approach (DSA) vs Posterior Approach (PA) in THA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17/0426
Record Dates: First submitted 2019-12-06; First posted 2019-12-10 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Surgery; Surgical Incision; Patient Satisfaction
Keywords: Total hip arthroplasty; Direct superior approach; Minimally invasive surgery; Implant position; Osteoarthritis; Posterior approach; Radiostereometric analysis
MeSH Terms: conditions — Surgical Wound; Patient Satisfaction; Osteoarthritis | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Direct Superior Approach (DSA) (Experimental): Direct superior incision during surgery
  Interventions: Device: Total hip arthroplasty
- Posterior Approach (PA) (Active Comparator): Posterior approach incision during surgery
  Interventions: Device: Total hip arthroplasty

INTERVENTIONS:
Device: Total hip arthroplasty — Surgical intervention designed to replace arthritic joint with artificial implant

SUMMARY:
Total Hip Arthroplasty (THA) is a highly effective treatment for patients with symptomatic hip osteoarthritis. The surgical approach in THA is important as it influences postoperative clinical recovery, functional outcomes, and implant positioning [1]. The evolution of surgical techniques in THA has led to the development of minimally invasive surgery, which is performed through smaller skin incisions, reduced soft tissue disruption and greater muscle preservation [2-10]. This prospective, randomised control study compares clinical and radiological outcomes in THA performed using the standard posterior approach (PA) and its less invasive modification, the direct superior approach (DSA). The study will include 80 patients with hip osteoarthritis undergoing THA. Following informed consent, patients will be randomised to one of the two treatment groups, and undergo THA using either the PA or DSA. The control group includes patients undergoing THA through the PA while the investigation group includes patients undergoing THA with the DSA. A further 25 patients randomly selected from each treatment group will undergo radiosteriometric analysis (RSA) to assess differences in early implant migration between PA and DSA groups.

Clinical and radiological outcomes of interest will be recorded by blinded observers at regular intervals for 2 years after surgery. The findings of this study will enable an improved understanding of differences in postoperative clinical recovery, functional outcomes, and implant positioning in THA performed using the DSA compared to the PA approach.

ELIGIBILITY:
Inclusion Criteria:

* Patient has hip osteoarthritis requiring primary THA

  * Patient and surgeon are in agreement that THA is the most appropriate treatment
  * Patient is fit for surgical intervention following review by surgeon and anaesthetist
  * Patient age: Patients 18-80 years of age inclusive
  * Gender: male and female
  * Patient must be capable of giving informed consent and agree to comply with the postoperative review program
  * Patient must be a permanent resident in an area accessible to the study site
  * Patient must have sufficient postoperative mobility to attend follow-up clinics and allow for radiographs to be taken

Exclusion Criteria:

* Patient is not suitable for primary THA e.g. patient requires revision surgery for previously failed THA

  * Patient is not medically fit for surgical intervention
  * Patients under the age of 18 or over 80 years of age
  * Patient is immobile or has another neurological condition affecting musculoskeletal function
  * Patient is already enrolled on another concurrent clinical trial
  * Patient is unable or unwilling to sign the informed consent form specific to this study
  * Patient is unable to attend the follow-up programme
  * Patient is non-resident in local area or expected to leave the catchment area postoperatively

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Pain in hip at 24 hours following surgery | 24 hours
  Pain at 24 hours following surgery as assessed using the visual analogue scale between patients undergoing PA for THA versus DSA for THA.

SECONDARY OUTCOMES:
Operating time | During the operation
  Operating time in minutes
Time to discharge | 6 weeks post operation
  Time to discharge in hours
Analgesia requirements | inpatient admission and postoperatively at 6 weeks, 6 months, 1 year and 2 years.
  Analgesia requirements
Oxford Hip Score (OHS) | Pre-op; 6 weeks post-op; 6 months post-op; 1 year post-op; 2 years post-op
  Patient recorded outcome measure via questionnaire. 48 is best score and 0 worst score
Hip injury and osteoarthritis outcome score (KOOS) | Pre-op; 6 weeks post-op; 6 months post-op; 1 year post-op; 2 years post-op
  Patient recorded outcome measure via questionnaire. 6 separate domains including pain, stiffness, quality of life, symptoms, and function; each domain creates percentage with overall cumulative percentage achieved; best score 100%
European Quality of Life questionnaire with 5 dimensions for adults (EQ-5D) | Pre-op; 6 weeks post-op; 6 months post-op; 1 year post-op; 2 years post-op
  Patient recorded outcome measure with 5 domains; score -1 to 1, with 1 being best score
Harris Hip Score [HHS] | Pre-op; 6 weeks post-op; 6 months post-op; 1 year post-op; 2 years post-op
  Patient recorded outcome measure via questionnaire. Scored 0-100 with 100 best possible outcome
Mobilisation distance | inpatient admission and postoperatively at 6 weeks, 6 months, 1 year and 2 years.
  Mobilisation distance in metres
Use of mobility aids | inpatient admission and postoperatively at 6 weeks, 6 months, 1 year and 2 years.
  Use of mobility aids
Femoral and acetabular implant early migration | postoperatively at 2 weeks, 6 weeks, 6 months, 1 year, and 2 years.
  Femoral and acetabular implant early migration as assessed using radiosteriometric analysis (RSA) This RSA will be performed on a cohort of 25 randomly selected patients from each treatment group.

CONTACTS AND LOCATIONS:
Locations (1):
- University College London Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plans

REFERENCES:
- [Derived] Kayani B, Konan S, Tahmassebi J, Ayuob A, Haddad FS. The direct superior approach versus posterior approach for total hip arthroplasty: study protocol for a prospective double-blinded randomised control trial. Trials. 2020 Jun 19;21(1):546. doi: 10.1186/s13063-020-04484-y. PMID 32560737